CLINICAL TRIAL: NCT02899182
Title: Mixture Nitrous Oxide - Oxygen 50-50% in Transrectal Prostate Biopsy Guided by Ultrasound
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Ismar Lima Cavalcanti, Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CAZARIMG
Record Dates: First submitted 2016-08-17; First posted 2016-09-14 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Nitrous Oxide; Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional group (Placebo Comparator): the conventional group (C) will receive local anesthesia at the puncture site plus inhalation of 100% oxygen a face mask.
  Interventions: Other: O2
- Nitrous Oxide NO (Experimental): The NO group receive local anesthesia at the puncture site plus inhalation N2O-O2 mixture by self-demand valve
  Interventions: Drug: Nitrous Oxide NO

INTERVENTIONS:
Drug: Nitrous Oxide NO — The NO group receive local anesthesia at the puncture site plus inhalation N2O-O2 mixture by self-demand valve
  Other Names: N2O
  Arms: Nitrous Oxide NO
Other: O2 — the conventional group (C) will receive local anesthesia at the puncture site plus inhalation of 100% oxygen a face mask.
  Other Names: conventional
  Arms: conventional group

SUMMARY:
Introduction: Transrectal ultrasound-guided prostate biopsy (TUPB) is the gold standard diagnostic tool for prostate cancer and, though may be well tolerated for some patients, about 65 to 90% of then still complain of discomfort, weather associated or not to pain. Therefore, as a manner of improvement in visual analogic pain score (VAS) and satisfaction between those patients, the aim of this study is to propose the gas mixture N2O-O2 50-50%, as a non-invasive, safe and cost-effective method to deliver analgesia and/or sedation, without the need for an anesthesiologist.

Materials and methods: A randomized clinical trial, simple blind, which took place in Hospital Universitário Antônio Pedro, Niteroi, RJ, within two groups containing 42 patients each, divided in conventional (C), which received 100% oxygen and nitrous oxide (NO), which received inhalation of the mixture N2O-O2 50-50% from a self-demand valve during exam. They were accessed for pain with VAS, answered a satisfaction task and were recorded about collateral side effects.

DETAILED DESCRIPTION:
Introduction:

Transrectal ultrasound-guided prostate biopsy (TUGP) is currently the gold standard method used for early cancer diagnosis of this gland, when associated with PSA plasma measurement. Although well tolerated by many patients, about 65-90% of men undergoing BPTU complain of discomfort, associated or not to pain. For better tolerance, various methods of analgesia and / or sedation have been proposed, such as nerve block periprostatic ( or intraprostatic, topical anesthesia with lidocaine or EMLA at the puncture site , general anesthesia with propofol and remifentanil and other invasive techniques.

Inhalation of N2O-O2 50-50% by self-demand valve proposed in this study can be a good alternative to invasive methods to be a safe technique, cost-effective, which promotes analgesia on demand, in order to increase the tolerance painful procedures as TUGP, regardless of the presence of anesthesiologists.

Nitrous oxide (N2O) can be self administered for analgesia in various procedures such as drug joint intra injections, vascular access puncture, flexible sigmoidoscopy and colonoscopy, ophthalmic procedures and prostate biopsy. In Europe it is used in emergencies in the care and transport accidents in ambulances.

The objective is to evaluate the efficiency of inhalation of N2O-O2 50-50% by self-demand valve, comparing it to a placebo group. In addition, investigators evaluated side events such as the adverse effects of administration of nitrous oxide to discuss their security procedures without the presence of anesthesiologist.

Materials and methods:

The trial will be done at Antonio Pedro University Hospital, Niterói, RJ - Brazil. Currently, the procedure is performed in the hospital outpatient clinics, without anesthesia.

Included patients are those undergoing transrectal prostate biopsy guided by ultrasound. Patients with failure to report the severity of the pain or unable to inhale through the device or Patients diagnosed with pulmonary hypertension, severe lung disease, or cardiac failure NYHA 3 and 4 will be excluded from the study The free and informed consent will be presented and signed by each volunteer participant, and the benefits of research clarified. 84 patients undergoing TUGP an outpatient will be randomized into two groups of 42. The conventional group (C) will receive local anesthesia at the puncture site plus inhalation of 100% oxygen a face mask (standard technique used routinely in our Hospital for this procedure). The NO group receive local anesthesia at the puncture site plus inhalation N2O-O2 mixture by self-demand valve An anesthesiologist will monitor the examinations respecting the resolution of the Federal Council of Medicine No. 1.802 / 2006, without being able to intervene in analgesia proposed by randomization. A visual analogy scale (VAS) pain 0-10 and a satisfaction form will be presented to the patient before the procedure and answered after it. The group will receive the mixture of N2O, O2 will be evaluated for the incidence of nausea, vomiting, dizziness, hemodynamic changes, fit of laughter and sleepiness during the examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing transrectal prostate biopsy guided by ultrasound

Exclusion Criteria:n.a

* Patients with failure to report the severity of the pain or unable to inhale through the device .
* Patients diagnosed with pulmonary hypertension , severe lung disease, or cardiac failure NYHA 3 and 4.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Pain reduction in patients undergoing transrectal ultrasound-guided prostate biopsy | 12 months
  Reduction on pain intensity evaluated by EVA scale

CONTACTS AND LOCATIONS:
Locations (1):
- Fluminense Federal University, Niterói, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No